CLINICAL TRIAL: NCT05546398
Title: SurveY Followed by a Retrospective Chart Review to Describe the Key Factors Leading to Physician's Decision to Treat Patients at High and Very High Cardiovascular Risk With hyperchOlesterolemia or Mixed Dyslipidemia With NUSTENDI® (Fixed Dose Combination of Bempedoic Acid 180mg and Ezetimibe 10mg) as add-on to Treatment With Maximally Tolerated Statin Therapy in Routine Clinical Practice
Brief Title: SurveY Followed by a Retrospective Chart Review to Describe the Key Factors Leading to Physician's Decision to Treat Patients at High and Very High Cardiovascular Risk With hyperchOlesterolemia or Mixed Dyslipidemia With NUSTENDI®
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Collaborators: Daiichi Sankyo Germany (Unknown)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: SYROS-DSE-BMP-01-21-EU
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Hypercholesterolemia; Mixed Dyslipidemia
Keywords: Hypercholesterolemia; Mixed dyslipidemia; NUSTENDI®; Statin therapy
MeSH Terms: conditions — Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Ezetimibe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physicians: Office-based cardiologists (OBCs) and lipid management specialists (LMSs) who are qualified for study participation regarding experience in lipid management therapy and treating a sufficient number of patients.
  Interventions: Other: No study drug
- High and Very High Cardiovascular Patients: Patients at high and very high cardiovascular risk as assessed by the office-based cardiologists and lipid management specialists with hypercholesterolemia or mixed dyslipidemia who received a prescription of bempedoic acid 180 mg fixed dose combination with ezetimibe 10 mg (FDC).
  Interventions: Drug: Bempedoic Acid 180Mg/Ezetimibe 10Mg Tab

INTERVENTIONS:
Drug: Bempedoic Acid 180Mg/Ezetimibe 10Mg Tab — No study drug was administered during this study.
  Other Names: NUSTENDI®
  Groups: High and Very High Cardiovascular Patients
Other: No study drug — No study drug was administered during this study.
  Groups: Physicians

SUMMARY:
In this study, a survey of office-based cardiologists and lipid management specialists will be conducted on treatment decisions for NUSTENDI® (bempedoic acid 180 mg fixed dose combination [FDC] with ezetimibe 10 mg) followed by a retrospective chart review of patients at high and very-high cardiovascular risk with hypercholesterolemia or mixed dyslipidemia who were treated with FDC as add-on to treatment with maximally tolerated statin therapy in routine clinical practice.

DETAILED DESCRIPTION:
The physician survey aims to understand the context of the real-world clinical setting and shed light on the utilization of FDC treatments by the prescribing physicians. The retrospective patient chart review will gain insights in real-world data of the patient's characteristics with a treatment decision for the FDC. No study drugs will be provided or administered as part of this protocol.

The objectives of the physician survey are the evaluation of the key factors for the therapy decision for the FDC:

* LDL-C levels at therapy decision and goal of LDL-C reduction
* Relevance of different factors and considerations
* Considerations of guidelines

The objectives of the retrospective patient chart review are to characterize the patients':

* Demographics
* LDL-C levels at therapy decisions
* Medical History
* Concomitant Diseases
* Lifestyle Modifications

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria for the office-based cardiologists and lipid management specialists are as follows:

  * More than 10 years of experience in medical practice
  * For office-based cardiologists: Supervision of at least 200 patients at high and very high cardiovascular risk as assessed by the office-based cardiologists with hypercholesterolemia or mixed dyslipidemia. For lipid management specialists: Supervision of at least 500 patients at high and very high cardiovascular risk as assessed by the lipid management specialists with hypercholesterolemia or mixed dyslipidemia
  * Working in practices to whom patients were either referred or had direct access to.
  * Availability to share medical files of consenting patients with study personnel (e.g. Clinical Research Associates) by remote quality review
  * At least 5 patients for the retrospective chart review

The inclusion criteria for the patients are as follows:

* Written informed consent to participate
* Patients at high and very high cardiovascular risk diagnosed with hypercholesterolemia or mixed dyslipidemia and treated with bempedoic acid 180 mg fixed dose combination with ezetimibe 10 mg (FDC) for at least 4 weeks at the discretion of the physician according to the German label

Exclusion Criteria:

* Any patient who did not meet all inclusion criteria noted above

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For the physician survey, office-based cardiologists and lipid management specialists must be qualified for study participation regarding experience in lipid management therapy and treating a sufficient number of patients. The office-based cardiologists and lipid management specialists will be preselected by the Medical Science Liaison Managers of DSDE.
  The retrospective patient chart review will include patients at high and very high cardiovascular risk as assessed by the office-based cardiologists and lipid management specialists with hypercholesterolemia or mixed dyslipidemia who received a prescription of FDC for at least 4 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Low density Lipoprotein-Cholesterol (LDL-C) Levels at Therapy Decision Based on Physician Survey | Up to 6 months
  Physicians will be surveyed to assess the LDL-C levels at the time of a therapy decision.
Reductions in Low density Lipoprotein-Cholesterol (LDL-C) Levels Based on Physician Survey | Up to 6 months
  Physicians will be surveyed to determine their anticipated reductions in LDL-C levels as a result of therapy.
Visual Analogue Scale (VAS) Score Evaluating Relevance of Decision Factors and Considerations Relevant to Therapy Decision Based on Physician Survey | Up to 6 months
  Physicians will be surveyed to determine the relevance of decision factors and considerations (including guidelines) that were relevant to their therapy decision based on a VAS ranging from 0 to 10.
Low density Lipoprotein-Cholesterol (LDL-C) Levels at Therapy Decision Based on a Retrospective Patient Chart Review | Up to 6 months
  A retrospective patient chart review will assess the LDL-C levels at the time of a therapy decision.
Number of Participants With Pre-specified Events in Their Medical History Based on a Retrospective Patient Chart Review | Up to 6 months
  A retrospective patient chart review will assess the number of participants with pre-specified events in their medical history.
Number of Participants With Specific Concomitant Diseases Based on a Retrospective Chart Review | Up to 6 months
  A retrospective patient chart review will assess the number of participants with specific concomitant diseases.
Number of Participants Implementing Specific Lifestyle Modifications Based on a Retrospective Patient Chart Review | Up to 6 months
  A retrospective patient chart review will assess the number of participants with specific lifestyle modifications.

CONTACTS AND LOCATIONS:
Locations (63):
- Germany (63):
  - Kardiologische Gemeinschaftspraxis (Bulut), Arnsberg
  - Dr. Georg Strack, Bad König
  - Dr. J. Nothroff, Berlin
  - Kardiologie am Spreebogen (Krackhardt), Berlin
  - Kardiologie Spreebogen Berlin (Haverkamp), Berlin
  - Kardiologische Facharztpraxis Winkelmann, Berlin
  - SPK-Studienzentrum Rankestraße GmbH, Berlin
  - Kardio Bonn, Bonn
  - Dr. Jaroslaw Sek, Chemnitz
  - Praxis Dipl.-med. Schermaul, Chemnitz
  - Praxis für Kardiologie und Schlafmedizin (Lichtenberg), Cologne
  - BAG Helmecke, Crivitz
  - Kardiologie Darmstadt, Darmstadt
  - MVZ Rhein-Main GmbH (Binder), Dreieich
  - Cardiologicum Dresden / Pirna (Hildebrandt), Dresden
  - Facharztzentrum Dresden-Neustadt GbR (Simonis), Dresden
  - PD Dr. Stephan Wiedemann, Dresden
  - Praxis Dr. Methfessel, Dresden
  - KardioPraxis Rote Straße (Stieber), Duisburg
  - Kardiologische Praxis (Warzok), Gotha
  - Kardiopraxis Greiz (Walter), Greiz
  - MVZ des Krankenhaus Greiz, Greiz
  - Kardiologie am Tibarg (Twisselmann), Hamburg
  - Diabetiker Zentrum Hannover (Fendler), Hanover
  - Kardiologie Haßloch (Gerhards), Haßloch
  - Kardiologie Alsterquelle, Henstedt-Ulzburg
  - Praxis Dr. Lißmann, Homburg
  - Gemeinschaftspraxis Dr. Täschner / Dr. Bonigut, Leipzig
  - Praxis Dr. Feige, Leipzig
  - Gemeinschaftspraxis Schauermann, Meiningen
  - Gemeinschaftspraxis Dres. med. Dittgen/Wilhelm/Rehlinger, Mettlach
  - Hausarztpraxis Doreen Drews, Michendorf
  - Hausarztpraxis Thorsten Drews, Michendorf
  - Kardio Praxis Mülheim (Möllenberg), Mülheim
  - Dres. Bettenworth & Partner, Münster
  - Gemeinschaftspraxis am Jahnufer (Schleß), Neu-Ulm
  - Kardiopraxis (Buchholz-Sanchez), Neustadt
  - Kardiologie am Weißen Turm (Stadelmann), Nuremberg
  - Praxis für Kardiologie (Laser), Nuremberg
  - Dres. Kornadt und Edel, Oberhausen
  - Praxis Dr. Spengler, Panitzsch
  - Kardiologische Praxis Papenburg Dr. Denchev, Papenburg
  - Kardiologische Praxis Papenburg Dr. Malazhavy, Papenburg
  - Kardiologische Praxis Papenburg Dr. Wilke, Papenburg
  - MVZ ambulantes Kardiologisches Zentrum Peine gGmbH, Peine
  - Kardiologe im MVZ Pfaffenhofen, Pfaffenhofen an der Ilm
  - Hausärztlich-Kardiologisches MVZ am Felsenkeller, Pirna
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci (Janßen), Potsdam
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci (Reibis), Potsdam
  - Nephrocare Püttlingen GmbH, Püttlingen
  - Praxisklinik Salzatal, Salzatal
  - Praxis Dr. Jax, Schwalmtal
  - Parkkardiologie (Wolf), Stahnsdorf
  - Parkkardiologie (Wuttke), Stahnsdorf
  - Praxis Dr. Birkenhagen, Stollberg
  - Kardiologische Gemeinschaftspraxis Dres. Klein & Neumann, Stuttgart
  - Studienzentrum der Herzklinik Ulm GbR, Ulm
  - Nephrologisches Zentrum Villingen Schwenningen (Hohenstein), Villingen-Schwenningen
  - Kardiologische Praxis (Elmas), Waghäusel
  - Praxis am Gutenbergplatz, Wiesbaden
  - Praxis Gerschanik, Wuppertal
  - Dres. Herrmann/Meyer/Teschner (Meyer), Würzburg
  - Praxis für Innere Medizin (Schwarz), Zwenkau

IPD SHARING:
Plan to Share IPD: No